CLINICAL TRIAL: NCT04802577
Title: The Level of Fatigue and Its Relationship With Disease Activity, Pain, Insomnia, and Psychometric Parameters in Primary Sjögren's Syndrome
Brief Title: Fatigue in Primary Sjögren's Syndrome
Status: Completed | Type: Observational
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Koray Ayar, Assistant Professor, Bursa Yuksek Ihtisas Training and Research Hospital
Other Study IDs: 2011-KAEK-25 2020/12-10
Record Dates: First submitted 2021-03-14; First posted 2021-03-17 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-11

CONDITIONS: Sjogren's Syndrome; Fatigue; Pain Syndrome; Depression; Anxiety; Fibromyalgia
MeSH Terms: conditions — Sjogren's Syndrome; Fatigue; Somatoform Disorders; Depression; Anxiety Disorders; Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Erythrocyte sedimentation rate, CRP, routine biochemical tests, and hemogram
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary Sjögren's syndrome: The patient's diagnosed with Primary Sjögren's according to 2016 ACR/EULAR classification criteria
  Interventions: Diagnostic Test: FACT-F questionnaire; Diagnostic Test: Beck Depression Inventory; Diagnostic Test: Beck Anxiety Inventory; Diagnostic Test: Insomnia severity index.; Other: ESSPRI; Other: ESSDAI; Other: Pain Detect Questionnaire
- Healthy Controls: Healthy hospital workers without any chronic disease
  Interventions: Diagnostic Test: FACT-F questionnaire; Diagnostic Test: Beck Depression Inventory; Diagnostic Test: Beck Anxiety Inventory; Diagnostic Test: Insomnia severity index.; Other: Pain Detect Questionnaire

INTERVENTIONS:
Diagnostic Test: FACT-F questionnaire — The questionnaire, based on patient report outcome data in which the presence of fatique is investigated in participants.
Diagnostic Test: Beck Depression Inventory — The questionnaire, based on patient report outcome data in which the presence of depression is investigated in participants.
Diagnostic Test: Beck Anxiety Inventory — The questionnaire, based on patient report outcome data in which the presence of anxiety is investigated in participants.
Diagnostic Test: Insomnia severity index. — The questionnaire, based on patient report outcome data in which the presence of insomnia is investigated in participants.
Other: ESSPRI — The questionnaire, based on patient report outcome data in which the severity of Sjögren's syndrome is investigated in participants.
  Groups: Primary Sjögren's syndrome
Other: ESSDAI — Activity scale in which the activity of Sjögren's syndrome is evaluated based on the laboratory and imaging tests of the patients and the examination findings of the evaluator.
  Groups: Primary Sjögren's syndrome
Other: Pain Detect Questionnaire — The questionnaire, based on patient report outcome data in which the severity and extent of pain in the body are investigated in participants.

SUMMARY:
Fatigue is a common clinical finding in Primary Sjögren's syndrome (PSS). In PSS, there is not enough data about the conditions in which fatigue develops and which clinical conditions the disease is associated with. This study was aimed to determine the level of fatigue in Primary Sjögren syndrome and to investigate the factors affecting the level of fatigue.

DETAILED DESCRIPTION:
While fatigue is seen with a prevalence of 7-8% in the normal population, it is more prevalent in Primary Sjögren's syndrome (PSS). In the studies conducted so far, the frequency of fatigue was seen at a frequency of over 30% in Primary Sjögren's syndrome. Although fatigue is so common in PSS, there is not enough data about the conditions in which fatigue develops in PSS. Other common conditions in PSS, apart from fatigue, are psychometric disorders such as common pain, depression and anxiety, and sleep disorders. In the studies conducted so far, each situation mentioned is common in PSS and seems to be related to each other. In the literature, there is no data on how many psychometric parameters, pain level, and insomnia affect fatigue and which are independent risk factors in PSS.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with PSS according to the 2016 ACR / EULAR criteria
* Healthy hospital staff

Exclusion Criteria:

* Pregnant women
* Cancer patients
* Those with other connective tissue diseases other than PSS
* Multiple sclerosis patients
* Chronic obstructive pulmonary disease
* Those with heart failure and adrenal insufficiency
* Those with renal failure: GFR <60 ml/min
* Anemia: Hemoglobin <11 g / dl in women, hemoglobin <12 g / dl in men
* Hypothyroidism: TSH >5 mu / L
* Those with electrolyte disturbance

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Volunteers who were followed up with a diagnosis of PSS in the center where the study was conducted and met the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
FACIT-F | day 1
  FUNCTIONAL ASSESSMENT OF CHRONIC ILLNESS THERAPY-FATİQUE

SECONDARY OUTCOMES:
BDI | day 1
  Beck Depression Inventory
BAI | day 1
  Beck Anxiety Inventory
ISS | day 1
  Insomnia Severity Scale
PDQ | day 1
  Pain Detect Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Koray Ayar, M.D., Principal Investigator — Univesity of Health Science, Bursa Yuksek Ihtisas Training and Research Hospital
Locations (1):
- Koray Ayar, Yıldırım, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No